CLINICAL TRIAL: NCT01022866
Title: Vancouver Falls Prevention Clinic Database
Brief Title: Falls Prevention Clinic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Other Study IDs: H09-02370
Record Dates: First submitted 2009-11-27; First posted 2009-12-01 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Falls
Keywords: falls; older adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
At the Falls Prevention Clinic, each subject receives a comprehensive assessment of his or her individual risk factors for falling in addition to a comprehensive medical examination. Recommendations and appropriate followup tests and referrals are ordered for patients on an individual basis.

Essential for medical advancement is the inquiry into information collected from medical records of older adults at high risk of falls and fracture. On such example is a retrospective chart review we conducted among patients who sustained a hip fracture [14]. The database we propose will provide novel insight into the identification of individuals at high risk for falls, key predictors of falls and associated mortality, morbidity, health related quality of life and healthcare resource utilization. In summary, our database will enable us to assess and improve quality of care, service delivery, patient outcomes, patient reported outcomes and track economic burden.

DETAILED DESCRIPTION:
Purpose: In community-dwelling seniors aged 70 years and older who attend the Vancouver Falls Prevention Clinic and who consent to allowing their data to form part of the Falls Prevention Clinic Database, we will audit charts to answer the following questions: 1) In terms of mobility and functional status, what characterizes the patient population that is referred to the Falls Prevention Clinic? 2) What is the physiological profile assessment (PPA) of individuals at the Falls Prevention Clinic? 3) What are the demographic characteristics? 4) What are factors that explain differences in health related quality of life and healthcare resource utilization? and 5) For individuals who have a high falls risk profile, what are their specific clinical outcome measures that indicate better or worse health related quality of life?

Objective: To develop a Falls Prevention Clinic Database for subjects who attend the Falls Prevention Clinic at Vancouver General Hospital and Lion's Gate Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥70 years attending a Falls Prevention Clinic Service;
* Understands, speaks, and reads English proficiently;
* MMSE [11] score > 24/30;
* A Physiological Profile Assessment (PPA) © [15] score of at least 2 SD above normal OR Timed Up and Go Test (TUG) 68 performance of greater than 15 seconds OR history of at least 2 falls in the previous 12 months;
* Expected to live greater than12 months;
* Living in the Metropolitan Vancouver area;
* Community-dwelling (i.e., not residing in a nursing home, extended care unit, or assisted-care facility);
* Able to walk 3 meters with or without an assistive device; and
* Able to provide written informed consent.

Exclusion Criteria:

* Diagnosed with a neurodegenerative disease (e.g., Parkinson's disease);
* Diagnosed with dementia (of any type);
* Had a stroke;
* Have clinically significant peripheral neuropathy or severe musculoskeletal or joint disease; or
* Have a history indicative of carotid sinus sensitivity (i.e., syncopal falls).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Falls Prevention Clinic
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Davis, Study Director — University of British Columbia; Karim Khan, Study Director — University of British Columbia; Teresa Liu-Ambrose, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Davis JC, Dian L, Khan KM, Bryan S, Marra CA, Hsu CL, Jacova P, Chiu BK, Liu-Ambrose T. Cognitive status is a determinant of health resource utilization among individuals with a history of falls: a 12-month prospective cohort study. Osteoporos Int. 2016 Mar;27(3):943-951. doi: 10.1007/s00198-015-3350-4. Epub 2015 Oct 8. PMID 26449355
- [Derived] Davis JC, Best JR, Bryan S, Li LC, Hsu CL, Gomez C, Vertes K, Liu-Ambrose T. Mobility Is a Key Predictor of Change in Well-Being Among Older Adults Who Experience Falls: Evidence From the Vancouver Falls Prevention Clinic Cohort. Arch Phys Med Rehabil. 2015 Sep;96(9):1634-40. doi: 10.1016/j.apmr.2015.02.033. Epub 2015 Apr 8. PMID 25862255
- [Derived] Davis JC, Bryan S, McLeod R, Rogers J, Khan K, Liu-Ambrose T. Exploration of the association between quality of life, assessed by the EQ-5D and ICECAP-O, and falls risk, cognitive function and daily function, in older adults with mobility impairments. BMC Geriatr. 2012 Oct 24;12:65. doi: 10.1186/1471-2318-12-65. PMID 23095570